CLINICAL TRIAL: NCT04613934
Title: Redesigning the Care Journey of Patients With Single-ventricle Congenital Heart Disease
Status: Completed | Type: Observational
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Carlos Miguel Mery, Associate Professor, University of Texas at Austin
Other Study IDs: 2019-08-0031
Record Dates: First submitted 2020-10-24; First posted 2020-11-03 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Single-ventricle; Congenital Heart Disease
Keywords: congenital heart disease; single-ventricle congenital heart disease; qualitative research; care experience
MeSH Terms: conditions — Univentricular Heart; Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this three-party collaboration, which includes The Texas Center for Pediatric and Congenital Heart Disease, the Value Institute for Health and Care, and the Design Institute for Health, all from University of Texas (UT) Dell Medical School, the investigators will explore how patient insights, data, storytelling, ideation, and prototyping can be employed to design a care delivery solution that enables patient outcome improvement. The goal of this project is to understand the life journey of patients with single-ventricle congenital heart disease and understand areas of that journey that can be improved. As such, the project intentionally does not start with a hypothesis, but instead seeks to gain insight of single-ventricle patients' care journey and based on that understanding identify opportunities for improvement.

DETAILED DESCRIPTION:
This collaborative research will utilize the Experience Group and Contextual Interview, two qualitative research methodologies, in order to understand and improve patients' and families with single-ventricle congenital heart disease (CHD) journey in care. There will be six main groups participating in the study: 1. Patients age 6 and older with a diagnosis of single-ventricle congenital heart disease; 2. Siblings (age 6 and older) of patients with single-ventricle CHD; 3. Parents or legal guardians of patients with single-ventricle CHD (regardless of patient age); 4. Pregnant parents who have a received a prenatal diagnosis of single-ventricle CHD; 5. Parents of deceased patients with single-ventricle CHD; 6. Adult partners of adult single-ventricle CHD patients.

Participants will take part in an Experience Group. The Experience Group methodology is a form of qualitative research that brings together a group of 4-8 people who share similar medical circumstances for a conversation. This methodology has been successfully used by researchers from the Value Institute for Health and Care to gain insights in different patient populations. The groups will take place at Dell Medical School, The Dell Pediatric Research Institute (across the street from Dell Children's Medical Center), or other convenient public location as needed to allow for the least amount of travel for participants. Each group lasts 60-90 minutes and encourages participants to discuss their conditions and experiences outside the hospital/clinic, specifically. Focusing on the lifestyle aspect of the patient experience enables insight into both the successes and the challenges faced outside the health care system and in unobservable situations. Conversation is encouraged by the facilitator, who offers topics such as "what makes a good/bad day?", "what are your aspirations, what are your fears?", and "what are some of the obstacles and burdens you face on a regular basis?" Using a research approach that employs semi-structured, open-ended questions directed towards the group as a whole, the investigators hope to learn about the unarticulated, unmet needs of these patients, both physical and emotional, and ranging both within and outside of the clinic. Participants will not be asked to take part in more than one Experience Group session. Due to the current COVID-19 pandemic, Experience Group sessions will be held virtually via Zoom.

Participants can elect to participate in a follow-up Contextual Interview following the Experience Groups. If the participants provide consent, they may be contacted for an interview. Not every patient that consents for participation will be asked to participate. Contextual Interviews will take place in participant's homes, or any other place of their choosing where they feel comfortable. Contextual Interviews will be performed by up to three personnel from the Design Institute for Health. The Design Institute has used this methodology extensively to identify needs and insights from patients to redesign care. Upon completion and approval of the optional model release part of the informed consent, audio recordings and photos may be taken. The Contextual Interviews do not follow a rigid question / answer scheme. Instead, their tone is conversational. Interview prompts will center around challenges the patients and families faced in their journey with CHD. Example questions may include, "When did you first receive the diagnosis?", "How do you feel about the care you were receiving?", "What, if anything, did the care team do to make you feel cared for?", "How did you feel about the location/environment?", and "What, if anything could have been different, improved or better for you?" Participants will not be asked to take part in more than one Contextual Interview session. Due to the current COVID-19 pandemic, Contextual Interviews will take place virtually via Zoom.

Finally, some participants will have the opportunity to take part in virtual workshops to discuss the challenges uncovered in the Experience Groups and Contextual Interviews and ideate potential solutions to such challenges. Workshops are ideation meetings lasting from a few hours to a full day and would include stakeholders from all three collaborators and patient and family representatives, if appropriate. Participants in workshops will be asked to comment on research insights, participate in ideation sessions (brainstorms), sketch and write up ideas and evaluate different service design concepts.

ELIGIBILITY:
Inclusion Criteria:

* Patients with any diagnosis of single-ventricle congenital heart disease, age 6 and older
* Parents or legal guardians of patients at any age with any diagnosis of single-ventricle congenital heart disease
* Siblings of patients with any diagnosis of single-ventricle congenital heart disease, age 6 and older
* Pregnant parents who have gotten any prenatal diagnosis of single-ventricle congenital heart disease
* Adult partners of adult patients with any diagnosis of single-ventricle congenital heart disease

Exclusion Criteria:

* Patients with a cognitive disability that prevents completion of the study procedures
* Patients, family members, and partners who do not speak English or Spanish

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients and families of patients with single-ventricle congenital heart disease
Sampling Method: Non-Probability Sample
Enrollment: 142 (Actual)
Dates: Start 2020-02-04 (Actual); Primary Completion 2020-10-16 (Actual); Study Completion 2020-10-16 (Actual)

PRIMARY OUTCOMES:
Identification of areas to be improved in patient and families' journey | 2 years
  This is a qualitative research study. The investigators are using a combination of Experience Group sessions, Contextual Interviews and workshops with patients and their family members to obtain information to identify areas of the lifelong journey of patient with single-ventricle congenital heart disease and their families that can be redesigned to improve the outcomes that matter most to the patients and their families

CONTACTS AND LOCATIONS:
Overall Officials: Carlos M Mery, MD, MPH, Principal Investigator — University of Texas at Austin
Locations (1):
- University of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mery CM, Well A, Taylor K, Carberry K, Colucci J, Ulack C, Zeiner A, Mizrahi M, Stewart E, Dillingham C, Cook T, Hartounian A, McCullum E, Affolter JT, Van Diest H, Lamari-Fisher A, Chang S, Wallace S, Teisberg E, Fraser CD Jr. Examining the Real-Life Journey of Individuals and Families Affected by Single-Ventricle Congenital Heart Disease. J Am Heart Assoc. 2023 Mar 7;12(5):e027556. doi: 10.1161/JAHA.122.027556. Epub 2023 Feb 21. PMID 36802928